CLINICAL TRIAL: NCT01012505
Title: The Effect of Exposure to Maternal Human Milk Odor on Physiological State of Preterms.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Dr. Ayala Maayan, Sheba Medical Cener
Other Study IDs: SHEBA-09-7392-AM-CTIL
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Health Preterm Infants With no Active Disease; Human Milk Nutrition; Incubator Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 20 preterm infants: 20 preterm infants without active disease
  Interventions: Other: adding pad with maternal milk in hte incubator

INTERVENTIONS:
Other: adding pad with maternal milk in hte incubator — 2 days prior to intervention - recording infants data and taking saliva cortisol adding pad with maternal milk - during 2 days - recording infants data and taking saliva cortisol.
  stopping intervention and for other 2 days recording infants data and taking saliva cortisol

SUMMARY:
Mammalian fetal sensory development comes in an invariant series, with the tactile/kinesthetic and chemosensory systems the earliest functioning and responsive to stimulation, implicating the importance of these foundational sensory systems for later development. Olfaction is essential for neonatal behavioral adaptation in many mammals, including humans. Experiments show that newborns recognize, and are soothed by, the smell of amniotic fluid. Provision of the mother's smell with breast pads, handkerchiefs she has worn, breast milk on a cotton ball or cotton applicator, or other means of providing odor and taste input can facilitate recognition by the infant's mother at a later time and does not appear to be detrimental to the stability of the infant.

Provision of the odor and taste of the mother's milk has been shown to facilitate the infant's mouthing, sucking, arousal, and calming from irritability, especially in preparation for oral feeding. Using 24 hour monitor analysis and cortisol saliva measurements, we will provide quantitive analysis to the effect of smell.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants at least 1 week of age
* no active disease or treatment (like respiratory support)
* place in incubator

Exclusion Criteria:

* active disease or treatment

Ages: 7 Days to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants at least 1 weekk of age no active disease or treatment (like respiratory support) place in incubator
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-12

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel